CLINICAL TRIAL: NCT01255540
Title: A Randomised Prospective Study of an Invasive Strategy Versus Medical Therapy in Patients Over 80 Years With Non ST-Elevation Myocardial Infarction (NSTEMI) or Unstable Angina Pectoris (UAP)
Brief Title: After Eighty Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Oslo University Hospital, Bjørn Bendz MD PhD, Oslo University Hospital
Other Study IDs: 08/326b
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease in patients over; 80 years of age.
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The rationale of the present clinical trial is to study whether an invasive strategy in clinical stable patients over 80 years with NSTEMI/UAP may improve rates of death, reinfarction, stroke, need of urgent revascularisation, myocardial function and quality of life. The invasive approach involves coronary angiography with immediate evaluation for three different treatment options; 1. Percutaneous coronary intervention (PCI), 2. Coronary artery bypass graft (CABG) or 3. medical treatment. Clinical practice shows that older patients are commonly treated less vigorously than younger patients and the present guidelines are based on a considerably younger population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years.
* Acute coronary syndrome (NSTEMI/UAP) with chest pain > 10 minutes, with or without ST-segment depression in ECG, and normal or elevated levels of troponin T or I. Elevated troponin levels are defined as values exceeding the 99 percentile of a normal population at the local laboratory at each participating site.
* Clinical stable

Exclusion Criteria:

* Age < 80 years.
* ST-segment elevation in ECG (STEMI)
* Clinical unstable with ongoing chest pain or other ischaemic symptoms/signs.
* Cardiogenic shock.
* Short life expectancy due to extra cardiac reason, ie. COPD, disseminated malignant disease, or other reason.
* Anamnestic indications for significant mental disorder, including dementia.
* Any condition which interferes with patients possibility to comply with protocol.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Multicenter study
Sampling Method: Probability Sample
Enrollment: 492 (Estimated)
Dates: Start 2010-12; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Composite endpoints. | One year follow up.
  Does an invasive strategy in clinical stable patients over 80 years with NSTEMI/UAP improve rates of death, reinfarction, stroke and need of urgent revascularisation?

SECONDARY OUTCOMES:
Death of any cause | One year from randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Derived] Berg ES, Tegn NK, Abdelnoor M, Roysland K, Ryalen PC, Aaberge L, Eek C, Oie E, Juliebo V, Gjertsen E, Ranhoff AH, Gullestad L, Nordstrand N, Bendz B; After Eighty Study Investigators. Long-Term Outcomes of Invasive vs Conservative Strategies for Older Patients With Non-ST-Segment Elevation Acute Coronary Syndromes. J Am Coll Cardiol. 2023 Nov 21;82(21):2021-2030. doi: 10.1016/j.jacc.2023.09.809. PMID 37968019
- [Derived] Tegn N, Eek C, Abdelnoor M, Aaberge L, Endresen K, Skardal R, Berg ES, Gullestad L, Bendz B. Patients aged 80 years or older with non-ST-elevation myocardial infarction or unstable angina pectoris randomised to an invasive versus conservative strategy: angiographic and procedural results from the After Eighty study. Open Heart. 2020 Jul;7(2):e001256. doi: 10.1136/openhrt-2020-001256. PMID 32719073
- [Derived] Tegn N, Abdelnoor M, Aaberge L, Hylen Ranhoff A, Endresen K, Gjertsen E, Skardal R, Gullestad L, Bendz B; After Eighty study investigators. Health-related quality of life in older patients with acute coronary syndrome randomised to an invasive or conservative strategy. The After Eighty randomised controlled trial. Age Ageing. 2018 Jan 1;47(1):42-47. doi: 10.1093/ageing/afx121. PMID 28985265
- [Derived] Tegn N, Abdelnoor M, Aaberge L, Endresen K, Smith P, Aakhus S, Gjertsen E, Dahl-Hofseth O, Ranhoff AH, Gullestad L, Bendz B; After Eighty study investigators. Invasive versus conservative strategy in patients aged 80 years or older with non-ST-elevation myocardial infarction or unstable angina pectoris (After Eighty study): an open-label randomised controlled trial. Lancet. 2016 Mar 12;387(10023):1057-1065. doi: 10.1016/S0140-6736(15)01166-6. Epub 2016 Jan 13. PMID 26794722